CLINICAL TRIAL: NCT03404466
Title: A Multicenter,Randomized,Open-label,Parallel-group,and Adaptive Design Clinical Study to Explore the Safety and Efficacy of Hypidone Hydrochloride Tablets in Treatment of Patients With Major Depressive Disorder
Brief Title: To Explore the Safety and Efficacy of Hypidone Hydrochloride Tablets in Treatment of Patients With MDD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Huahai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYP201-CTP
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group one (Experimental): 10 mg of Hypidone Hydrochloride tablets
  Interventions: Drug: Hypidone Hydrochloride tablets
- experimental group two (Experimental): 20 mg of Hypidone Hydrochloride tablets
  Interventions: Drug: Hypidone Hydrochloride tablets

INTERVENTIONS:
Drug: Hypidone Hydrochloride tablets — Hypidone Hydrochloride tablets 10 or 20mg/day Study drug is to be given orally, twice daily, for 6 weeks

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Hypidone Hydrochloride tablets in treatment of patients with major depressive disorder (MDD) by evaluating the change of MADRS total score from baseline to week 6.

DETAILED DESCRIPTION:
A total of 40 major depressive disorder (MDD) subjects between the ages of 18-65 who have current major depressive disorder diagnosed by DSM-5 will be recruited, Subjects will be accepted into the protocol after an opportunity to review and provide voluntary written informed consent and completion of a comprehensive medical and psychiatric history, physical examination, mental status examination, and routine laboratory assessments The subjects will accept the drug treatment twice daily orally for 6 weeks, During the treatment follow up will occur at 8±1 days after treatment, 15±1 days after treatment, 29±2 days after treatment ,43±2 days after treatment to evaluate the safety and efficacy of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, 18-65 years old, Male or female
2. Current major depressive disorder diagnosed by DSM-5,single episode(296.21, 296.22, 296.23),or recurrent episode(296.31, 296.32, 296.33)
3. Montgomery-Åsberg Depression Rating Scale (MADRS) total scores in both Screening and Baseline ≥ 26
4. The first item of MADRS in both Screening and Baseline ≥ 3
5. CGI-S in both Screening and Baseline ≥ 4
6. Able to provide written informed consent

Exclusion Criteria:

1. Patients accord with other mental disorders diagnosed by DSM-5
2. Attempts to suicide, or who presently have a high risk of suicide, or The tenth item (Suicidal ideation) of C-SSRS ≥ 3
3. Baseline total scores compared with the screening period, the reduction rate of MADRS ≥ 25%
4. Subjects with serious or uncontrolled cardiovascular disease, liver disease, kidney disease, blood disease, endocrine disease, respiratory disease
5. Subjects with clinically significant ECG abnormal(Male QTcF ≥ 450 msec, Female QTcF ≥ 470 msec )
6. Treatment with a MAOI within the 2 weeks prior to the first dose of trial medication
7. practicing 2 different treatment methods of antidepressants as recommended dose of full course
8. Subjects who have had a Vagus Nerve Stimulation(VNS) device implanted or who have received Modified Electric Convulsive Therapy(MECT) or Transcranial Magnetic Stimulation (TMS) within 3 months of Screening, received light treatment, laser treatment, acupuncture and other Chinese medicine treatment, biofeedback treatment within 2 weeks of Screening
9. Subjects with a history of true allergic response to more than 1 class of medications
10. Subjects who participated in a clinical trial within the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-02-24 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Screening,Baseline,8 day after treatment,15 day after treatment,29 day after treatment,43 day after treatment
  Change from baseline in MADRS scores，the *total* score ranges[0,60],higher values represent a worse outcome

SECONDARY OUTCOMES:
Change in Hamilton Depression Scale 17 items(HAMD17) | Baseline,8 day after treatment,15 day after treatment,29 day after treatment,43 day after treatment
  Change from baseline in HAMD17 scores,the *total* score ranges[0,50],higher values represent a worse outcome
Change in Hamilton Anxiety Rating Scale (HAM-A) | Baseline, 8 day after treatment,15 day after treatment,29 day after treatment ,43 day after treatment
  Change from baseline in HAM-A scores,the *total* score ranges[0,56],higher values represent a worse outcome
Change in Clinical Global Impression of Severity Scale(CGI-S) | Screening,Baseline, 8 day after treatment,15 day after treatment,29 day after treatment,43 day after treatment
  Change from baseline in CGI-S scores,the *total* score ranges[0,7],higher values represent a worse outcome
Change in Clinical Global Impression of Improvement Scale(CGI-I) | 8 day after treatment,15 day after treatment,29 day after treatment,43 day after treatment
  the *total* score ranges[0,7],higher values represent a worse outcome
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline,15 day after treatment,43 day after treatment
  Safety index，no total score

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai mental health center, Shanghai, Shanghai Municipality, China